CLINICAL TRIAL: NCT05490563
Title: A Double-blind, Randomized, Placebo Controlled, Trial to Assess Safety and Efficacy of SLS-005 (Trehalose Injection, 90.5 mg/mL for Intravenous Infusion) for the Treatment of Adults With Spinocerebellar Ataxia
Brief Title: STRIDES - a Clinical Research Study of an Investigational New Drug to Treat Spinocerebellar Ataxia
Acronym: STRIDES
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: This was a business decision due to financial considerations, not based on data related to safety or therapeutic effects.
Sponsor: Seelos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SLS-005-302
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Spinocerebellar Ataxia Type 3
MeSH Terms: conditions — Machado-Joseph Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SLS-005 0.75 g/kg Dose (Experimental): SLS-005 (trehalose injection, 90.5 mg/mL for intravenous infusion). SLS-005 will be administered as a weight-based dose of 0.75 g/kg by IV infusion once a week.
  For 52 weeks
  Interventions: Drug: SLS-005
- SLS-005 0.50 g/kg Dose (Experimental): SLS-005 (trehalose injection, 90.5 mg/mL for intravenous infusion). SLS-005 will be administered as a weight-based dose of 0.50 g/kg by IV infusion once a week.
  For 52 weeks
  Interventions: Drug: SLS-005
- Placebo volume equivalent to a SLS-005 0.75 g/kg dose calculation (Placebo Comparator): Placebo (sodium chloride injection, 0.9, USP) will be administered by IV infusion once a week as a weight-based volume equivalent to a SLS-005 0.75 g/kg dose.
  For 52 weeks
  Interventions: Drug: Placebo
- Placebo volume equivalent to a SLS-005 0.50 g/kg dose calculation (Placebo Comparator): Placebo (sodium chloride injection, 0.9, USP) will be administered by IV infusion once a week as a weight-based volume equivalent to a SLS-005 0.50 g/kg dose.
  For 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SLS-005 — SLS-005
  Arms: SLS-005 0.50 g/kg Dose; SLS-005 0.75 g/kg Dose
Drug: Placebo — Placebo (sodium chloride injection, 0.9%, USP)
  Arms: Placebo volume equivalent to a SLS-005 0.50 g/kg dose calculation; Placebo volume equivalent to a SLS-005 0.75 g/kg dose calculation

SUMMARY:
Phase 2b/3 double blind, randomized, placebo-controlled trial to assess safety and efficacy of SLS-005 (trehalose injection, 90.5 mg/mL for intravenous infusion) for the treatment of adults with spinocerebellar ataxia).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled trial to assess the safety and efficacy of SLS-005 for the treatment of adults with SCA. The study consists of a 2-week screening period, a 52-week treatment period, and a 2-week safety follow-up period. Eligible participants between the ages of 18-75 years, will be randomized to treatment with SLS-005 or equivalent placebo (sodium chloride injection, 0.9%, USP). The study plans to enroll up to 245 participants with SCA3.

Biomarkers associated with neuro-axonal injury, pharmacokinetics, Modified Scale for Assessment and Rating of Ataxia (m-SARA), Clinical Global Impression of Severity (CGI-S), Patient Global Impression of Severity (PGI-S), and Friedreich's Ataxia Rating Scale - Activities of Daily Living (FARS-ADL), will be assessed at screening and/or baseline and at scheduled times throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Men and women, 18 to 75 years (inclusive) of age.
3. Clinical diagnosis of SCA3 with documented genetic confirmation.
4. m-SARA total score ≥ 4 at the screening visit.
5. m-SARA gait component score ≥ 1 at the screening visit.
6. Body Mass Index (BMI) between 18 kg/m2 and 35 kg/m2 (inclusive).
7. Stable doses of all concomitant medications for at least 30 days prior to the screening visit.
8. Negative serum beta-human chorionic gonadotropin (ß-hCG) pregnancy result at the screening visit for female participants of childbearing potential.
9. Willingness to comply with sexual abstinence or contraception guidelines of this study.

Exclusion Criteria:

1. Any hereditary ataxia that is not genetically confirmed to be SCA type 3, or any type of ataxia that is acquired or secondary to another medical condition including but not limited to, alcoholism, head injury, multiple sclerosis, olivopontocerebellar atrophy, multiple system atrophy, or stroke.
2. A score of 4 on any 1 of the 4 items that comprise the m-SARA.
3. Current participation in another clinical trial or completed participation in an interventional trial less than 30 days prior to the screening visit (90 days for a biological treatment).
4. Current diagnosis and/or healthcare professional-recommended treatment (medication and/or diet) of diabetes mellitus type 1 or type 2.
5. Hemoglobin A1c (HbA1c) ≥ 6.5% at the screening visit
6. Prior treatment with SLS-005, any other IV trehalose formulation, or known hypersensitivity to trehalose.
7. Pregnant or breastfeeding.
8. History of alcohol or drug abuse within the last 2 years.
9. Chronic liver disease including Hepatitis B; Hepatitis C unless successful curative treatment is documented; human immunodeficiency virus (HIV) infection.
10. Prior history of drug-induced liver injury (DILI) and/or laboratory results at screening that indicate inadequate liver function (e.g., alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyl transferase [GGT] > 2 times the upper limit of normal [x ULN] and/or total bilirubin level > 2 x ULN).
11. Laboratory results at screening that indicate inadequate renal function (e.g., estimated creatinine clearance of < 60 mL/min calculated by the Cockcroft and Gault formula).
12. Any current cardiovascular disease or abnormality on 12-lead ECG at screening that, in the investigator's opinion, is clinically significant and could be a potential safety risk to the participant.
13. Any current psychiatric, neurological, or cognitive disorder that, in the investigator's opinion, may interfere with the participant's ability to provide informed consent or appropriately complete the study's safety or efficacy assessments.
14. Significant suicide risk as indicated by a "yes" response to question #4 or #5 under Suicidal Ideation in the past 6 months or any "yes" response under Suicidal Behavior in the past 3 years on the Columbia Suicide Severity Rating Scale (C-SSRS) during the screening visit.
15. Any other medical condition or abnormal finding during screening that, in the investigator's opinion, could confound collection or interpretation of safety or efficacy data or be a potential safety risk to the participant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy: m-SARA | 52 weeks
  Mean change from baseline in Modified Scale for Assessment and Rating of Ataxia (m-SARA) total score at week 52

SECONDARY OUTCOMES:
Efficacy: CGI-S | 4, 13, 26, 39, and 52 weeks
  Mean change from baseline in Clinical Global Impression of Severity (CGI-S) score at week 52
Efficacy: PGI-S | 4, 13, 26, 39, and 52 weeks
  Mean change from baseline in Patient Global Impression of Severity (PGI-S) score at week 52
Efficacy: FARS-ADL | 4, 13, 26, 39, and 52 weeks
  Mean change from baseline in Friedreich's Ataxia Rating Scale (FARS) for the assessment of performance in basic activities that are typically required daily for independent living.
Efficacy: m-SARA | 26 weeks
  Mean change from baseline in m-SARA total score at week 26.
Efficacy: m-SARA | 52 weeks
  Mean change from baseline in m-SARA total score at weeks 4, 13, 26, 39, and 52
Safety: Adverse Events | 56 weeks
  Incidences of Treatment-Emergent Adverse Events and Serious Adverse Events (SAEs), including clinically significant laboratory and electrocardiogram (ECG) abnormalities.

CONTACTS AND LOCATIONS:
Locations (23):
- United States (7):
  - UCLA, Los Angeles, California
  - UCHealth Neurosciences Center - Anschutz Medical Campus, Aurora, Colorado
  - University of South Florida, Tampa, Florida
  - Harvard Medical School - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - UT Southwestern Medical Center, Dallas, Texas
  - Swedish Neuroscience Specialists - Movement Disorders, Seattle, Washington
- The Alfred Hospital, Melbourne, Victoria, Australia
- Brazil (3):
  - Hospital de Clinicas de Porto Alegre UFRGs, Porto Alegre, Rio Grande do Sul
  - Policlinica - Universidade Estadual de Campinas UNICAMP, Campinas, São Paulo
  - University of Sao Paulo, Ribeirão Preto, São Paulo
- Germany (2):
  - University Hospital of Leipzig, Leipzig, Saxony
  - Department of Neurology and Hertie Institute for Clinical Brain Research, Tübingen
- Portugal (3):
  - Centro Hospitalar e Universitrio de Coimbra, Coimbra
  - Hospital de Santa Maria, Centro Hospitalar Lisboa Norte, Neurologia, Lisbon
  - Hospital de Santo António, Centro Hospitalar Universitário do Porto, Porto
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center/Sungkyunwhan Universtiy School of Medicine, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Fe, Valencia
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No